CLINICAL TRIAL: NCT07303218
Title: The HER Project: Homologous Recombination Deficiency in EGFR-Mutated NSCLC, a Retrospective and Prospective Translational Single-center Study
Brief Title: The HER Project: HRD in EGFR-mutated NSCLC
Acronym: HER
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Francesca Rita Ogliari, Medical Doctor, IRCCS San Raffaele
Other Study IDs: The HER Project
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: EGFR; Non Small Cell Lung Cancer; Homologous Recombination Deficiency; PARP Inhibitor
Keywords: EGFR; Non small cell lung cancer; NSCLC; Homologous Recombination Deficiency; HRD; PARP Inhibitors; cell lines; organoids; Osimertinib; Olaparib; Genomic Scarring Score; TP53
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tumor samples (biopsies, surgical samples)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective Cohort: Patients with metastatic EGFR-mutated NSCLC diagnosed and treated between January 2020 and September 2025, with tumour tissue available for HRD analysis.
  Interventions: Other: No Intervention: Observational Cohort
- Prospective Cohort: Patients with newly diagnosed metastatic EGFR-mutated NSCLC, with baseline tumour tissue available for HRD testing and prospectively collected clinical follow-up.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — Observational study only; participants receive standard-of-care treatments not assigned by the study

SUMMARY:
This observational retrospective-prospective study aims to evaluate the prevalence of homologous recombination deficiency (HRD) in metastatic EGFR mutated NSCLC and to assess its correlation with clinical and molecular features. Based on the hypothesis that HRD identifies a distinct EGFRm subgroup with prognostic value and a potential sensitivity to PARP inhibitor-based strategies, translational analysis will be performed with multiple pre-clinical models, ranging from human cancer cells to murine models.

DETAILED DESCRIPTION:
Introduction

Lung cancer is the most common diagnosed cancer, with almost 2.5 million new cases per year, and the leading cause of cancer-related death (18.7%), according to GLOBOCAN (2022). Non-small cell lung cancer (NSCLC) is the most prevalent subtype, accounting for 85% of lung cancers. Epidermal growth factor receptor (EGFR) is a transmembrane tyrosine kinase receptor that regulates survival, proliferation and differentiation in mammalian cells. EGFR mutations occur in around 30% of patients affected by NSCLC, representing the second most frequent targetable oncogenic driver in NSCLC.

The treatment landscape for metastatic EGFR-mutated (EGFRm) NSCLC has significantly evolved since the introduction of 1st generation tyrosine kinase inhibitors (TKIs) in 2010. While osimertinib (a 3rd generation TKI) is currently the standard first-line treatment worldwide in the advanced setting, emerging combination strategies, such as osimertinib plus chemotherapy (FLAURA2 trial) or lazertinib plus amivantamab (MARIPOSA trial), improved progression-free survival (PFS) and overall survival (OS) compared to TKI alone. However, these drug combinations often cause increased treatment-related toxicities, impacting both patients' quality of life and healthcare costs. For this reason, it becomes crucial to identify predictive biomarkers to guide patient selection for combination therapies. For example, post-hoc analyses of FLAURA2 were conducted on poor-risk populations, such as EGFRm patients with high tumour burden or TP53 co-mutations. Despite better outcomes of chemotherapy plus osimertinib across all patient subgroups, only 1 out of 4 patients had baseline tissue samples available for wider genome sequencing. Therefore, understanding the role of co-alterations in EGFRm tumours remains to be explored, particularly those associated with shorter OS and/or more aggressive clinical presentations.

Targeting HRD pathway with PARP-inhibitors in Non-small cell lung cancer

Homologous recombination deficiency (HRD) is a condition linked to an impaired DNA repair mechanism that contributes to genomic instability in several cancers, including NSCLC. PARP-inhibitors (PARPi), drugs targeting a key protein involved in DNA repair, are already available in clinical practice for the treatment of other HRD-positive subgroups of solid tumours (e.g. breast, ovarian, prostate cancer). In NSCLC, however, their clinical benefit remains unclear. Previous studies evaluating PARPi in NSCLC, including combinations with chemotherapy or immunotherapy, have shown modest or non-significant improvements in PFS and OS. However, a significant limitation of these studies is the lack of HRD status assessment, which may have diluted the expected benefits in HRD-positive patients.

Interestingly, emerging evidence suggests that a higher Genomic Scarring Score (GSS), a surrogate for HRD, may predict PARPi sensitivity better than the traditional assessment of the mutational status of homologous recombination repair (HRR) genes. In this study, the administration of PARPi significantly delayed tumour growth in patient-derived xenograft (PDXs) with high GSS, half of which carried pathogenic/likely pathogenic somatic HRR mutations. Importantly, favourable responses to the PARPi-olaparib were observed regardless of HRR gene mutation status, underscoring the potential of GSS as a robust biomarker to more effectively select patients for PARPi-based therapies.

HRD in EGFR mutated NSCLC

In a Chinese cohort of HRD-positive NSCLC, EGFR-mutated tumours are associated with poor TKI response, which might be explained by gene amplifications like MET, a common resistance mechanism that can be promoted by HRD. Studies also showed the co-occurrence of biallelic TP53 mutations and high HRD score in poor-risk EGFRm NSCLC, suggesting a link between this tumour genotype and TKI-resistance. In preclinical models of NSCLC, osimertinib-resistant EGFRm cell lines exhibited sensitivity to olaparib, leading to increased DNA damage and cell death via a pro-oxidant state. Moreover, combining osimertinib with a PARPi in vivo significantly improved tumour regression compared to osimertinib alone. Altogether, these findings lead to hypothesize that the HRD positive score/GSS may define a patient subgroup that could benefit from PARPi-based combination therapy.

Clinical trials evaluating EGFR-TKIs with PARPi failed to achieve their primary endpoint of PFS, possibly due to a lack of patient selection based on HRD score or other molecular criteria. However, subsequent analyses of the GOAL trial found a stronger synergy between gefitinib (a 1st generation TKI) and olaparib in tumours with higher BRCA1 expression, supporting a predictive role for targeting DNA damage repair pathways. In operable NSCLCs, the percentage of HRD positive tumours is ~20-30%, suggesting that the acquisition of HRD status could be an early event. Importantly, a similar incidence was observed in a Chinese cohort of any-stage EGFRm or ALK-rearranged NSCLC patients in which the cases with high HRD score are ~33% of the total. The sensitivity of EGFRm tumours to platinum-based doublets, which is a known characteristic of HRD-positive tumours, and a larger compendium evidence of chromosomal instability further support exploring the role of HRD in EGFR-mutated lung cancer, paving the way for new targeted therapeutic approaches.

The HER Project

With the HER project, we will investigate the role of HRD and genomic instability (GSS) in EGFRm NSCLC by i) defining the fraction of metastatic EGFRm tumours with HRD positive score, ii) correlating HRD score with patient outcomes, and iii) assessing the synergic efficacy of EGFR-TKIs plus PARPi based on the HRD score in different preclinical settings, ranging from cell lines to a murine model of spontaneous EGFRm lung cancer. We expect that this drug combination will be effective in a specific subset of EGFR tumors. However, even if we won't observe any relevant findings by targeting this pathway, our work will increase our knowledge about DNA damage repair and drug resistance in EGFRm tumours.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for participation in the study. However, since a part of the study is retrospective and, considering the large sample sizes required and considering that the disease involved in this study affects elderly subjects with co-morbidities and presents a significant mortality rate based on the stage of the disease, deceased and untraceable patients will also be included.
2. Age ≥18 years old
3. Have a metastatic histologically confirmed NSCLC
4. Presence of EGFR common mutations (i.e. ex19del and L858R)
5. Have sufficient biological material to assess genomic profiling with AmoyDx Focus panel or similar
6. Clinical data available

Exclusion Criteria:

1. Insufficient baseline tumour tissue (unsuitable for HRD scoring)
2. Presence of EGFR uncommon mutations (i.e. ex20ins)
3. Known presence of co-occurring uncommon EGFRm, ALK, ROS1, or other main oncogenic drivers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with metastatic EGFR-mutated NSCLC eligible for treatment with EGFR-TKI according to standard clinical practice, with available tumor tissue suitable for HRD testing
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HRD in metastatic EGFRm NSCLC | Baseline (T0), on diagnostic tumour sample
  Proportion of EGFRm NSCLC with an HRD positive score evaluated by AmoyDx HRD Panel or similar (GSS ≥ 50).

SECONDARY OUTCOMES:
Correlation between HRD status and clinical outcomes and molecular features | Up to 3 years of follow-up for PFS/OS; baseline for clinical and molecular characteristics.
  Assessment of the association between HRD status (positive vs negative) and:
  * Clinical outcomes including progression-free survival (PFS), defined as time from initiation of first line treatment to evidence of progressive disease, and overall survival (OS), defined as time from initiation of first line treatment to death.
  * Baseline clinical characteristics
  * Baseline molecular features including EGFR mutation type, variant allele frequency (VAF) and other co-occurring molecular alterations

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Rita Ogliari, Medical Doctor, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- Dept. Medical Oncology, Milan, MI, Italy

REFERENCES:
- [Background] Drews RM, Hernando B, Tarabichi M, Haase K, Lesluyes T, Smith PS, Morrill Gavarro L, Couturier DL, Liu L, Schneider M, Brenton JD, Van Loo P, Macintyre G, Markowetz F. A pan-cancer compendium of chromosomal instability. Nature. 2022 Jun;606(7916):976-983. doi: 10.1038/s41586-022-04789-9. Epub 2022 Jun 15. PMID 35705807
- [Background] Fang S, Wang Z, Guo J, Liu J, Li C, Liu L, Shi H, Liu L, Li H, Xie C, Zhang X, Sun W, Li M. Correlation between EGFR mutation status and response to first-line platinum-based chemotherapy in patients with advanced non-small cell lung cancer. Onco Targets Ther. 2014 Jul 1;7:1185-93. doi: 10.2147/OTT.S63665. eCollection 2014. PMID 25061320
- [Background] Klinakis, A. et al. 1277P HRD status of patients with early stage non-small cell lung cancer. Annals of Oncology 34, S737-S738 (2023)
- [Background] Karachaliou N, Arrieta O, Gimenez-Capitan A, Aldeguer E, Drozdowskyj A, Chaib I, Reguart N, Garcia-Campelo R, Chen JH, Molina-Vila MA, Rosell R; Spanish Lung Cancer Group (SLCG). BRCA1 Expression and Outcome in Patients With EGFR-Mutant NSCLC Treated With Gefitinib Alone or in Combination With Olaparib. JTO Clin Res Rep. 2020 Oct 23;2(3):100113. doi: 10.1016/j.jtocrr.2020.100113. eCollection 2021 Mar. PMID 34589994
- [Background] Garcia-Campelo R, Arrieta O, Massuti B, Rodriguez-Abreu D, Granados ALO, Majem M, Vicente D, Lianes P, Bosch-Barrera J, Insa A, Domine M, Reguart N, Guirado M, Sala MA, Vazquez-Estevez S, Caro RB, Drozdowskyj A, Verdu A, Karachaliou N, Molina-Vila MA, Rosell R; Spanish Lung Cancer Group (SLCG). Combination of gefitinib and olaparib versus gefitinib alone in EGFR mutant non-small-cell lung cancer (NSCLC): A multicenter, randomized phase II study (GOAL). Lung Cancer. 2020 Dec;150:62-69. doi: 10.1016/j.lungcan.2020.09.018. Epub 2020 Oct 3. PMID 33070053
- [Background] Marcar L, Bardhan K, Gheorghiu L, Dinkelborg P, Pfaffle H, Liu Q, Wang M, Piotrowska Z, Sequist LV, Borgmann K, Settleman JE, Engelman JA, Hata AN, Willers H. Acquired Resistance of EGFR-Mutated Lung Cancer to Tyrosine Kinase Inhibitor Treatment Promotes PARP Inhibitor Sensitivity. Cell Rep. 2019 Jun 18;27(12):3422-3432.e4. doi: 10.1016/j.celrep.2019.05.058. PMID 31216465
- [Background] Feng J, Lan Y, Liu F, Yuan Y, Ge J, Wei S, Luo H, Li J, Luo T, Bian X. Combination of genomic instability score and TP53 status for prognosis prediction in lung adenocarcinoma. NPJ Precis Oncol. 2023 Oct 31;7(1):110. doi: 10.1038/s41698-023-00465-x. PMID 37907595
- [Background] Fischer A, Bankel L, Hiltbrunner S, Rechsteiner M, Ruschoff JH, Rushing EJ, Britschgi C, Curioni-Fontecedro A. Mutational Landscape and Expression of PD-L1 in Patients with Non-Small Cell Lung Cancer Harboring Genomic Alterations of the MET gene. Target Oncol. 2022 Nov;17(6):683-694. doi: 10.1007/s11523-022-00918-6. Epub 2022 Sep 22. PMID 36136211
- [Background] Wang Y, Ma Y, He L, Du J, Li X, Jiao P, Wu X, Xu X, Zhou W, Yang L, Di J, Zhu C, Xu L, Sun T, Li L, Liu D, Wang Z. Clinical and molecular significance of homologous recombination deficiency positive non-small cell lung cancer in Chinese population: An integrated genomic and transcriptional analysis. Chin J Cancer Res. 2024 Jun 30;36(3):282-297. doi: 10.21147/j.issn.1000-9604.2024.03.05. PMID 38988485
- [Background] Tsilingiri K, Chalari A, Christopoulou G, Voutsina A, Constantoulakis P, Potaris Kappa, Vamvakaris I, Hatzidaki D, Zachou G, Vatsellas G, Georgoulias V, Kotsakis A, Klinakis A. Genomic scarring score predicts the response to PARP inhibitors in non-small cell lung cancer. NPJ Precis Oncol. 2024 Dec 26;8(1):291. doi: 10.1038/s41698-024-00777-6. PMID 39725687
- [Background] Clarke JM, Patel JD, Robert F, Kio EA, Thara E, Ross Camidge D, Dunbar M, Nuthalapati S, Dinh MH, Bach BA. Veliparib and nivolumab in combination with platinum doublet chemotherapy in patients with metastatic or advanced non-small cell lung cancer: A phase 1 dose escalation study. Lung Cancer. 2021 Nov;161:180-188. doi: 10.1016/j.lungcan.2021.09.004. Epub 2021 Sep 17. PMID 34607210
- [Background] Ahn MJ, Bondarenko I, Kalinka E, Cho BC, Sugawara S, Galffy G, Shim BY, Kislov N, Nagarkar R, Demedts I, Gans SJM, Mendoza Oliva D, Stewart R, Lai Z, Mann H, Shi X, Hussein M. Durvalumab in Combination With Olaparib Versus Durvalumab Alone as Maintenance Therapy in Metastatic NSCLC: The Phase 2 ORION Study. J Thorac Oncol. 2023 Nov;18(11):1594-1606. doi: 10.1016/j.jtho.2023.06.013. Epub 2023 Jun 29. PMID 37390980
- [Background] Ramalingam SS, Thara E, Awad MM, Dowlati A, Haque B, Stinchcombe TE, Dy GK, Spigel DR, Lu S, Iyer Singh N, Tang Y, Teslenko I, Iannotti N. JASPER: Phase 2 trial of first-line niraparib plus pembrolizumab in patients with advanced non-small cell lung cancer. Cancer. 2022 Jan 1;128(1):65-74. doi: 10.1002/cncr.33885. Epub 2021 Sep 3. PMID 34478166
- [Background] Hochmair M, Schenker M, Cobo Dols M, Kim TM, Ozyilkan O, Smagina M, Leonova V, Kato T, Fedenko A, De Angelis F, Rittmeyer A, Gray JE, Greystoke A, Aggarwal H, Huang Q, Zhao B, Lara-Guerra H, Nadal E. Pembrolizumab With or Without Maintenance Olaparib for Metastatic Squamous NSCLC That Responded to First-Line Pembrolizumab Plus Chemotherapy. J Thorac Oncol. 2025 Feb;20(2):203-218. doi: 10.1016/j.jtho.2024.10.012. Epub 2024 Oct 28. PMID 39477187
- [Background] Fennell DA, Porter C, Lester J, Danson S, Blackhall F, Nicolson M, Nixon L, Gardner G, White A, Griffiths G, Casbard A. Olaparib maintenance versus placebo monotherapy in patients with advanced non-small cell lung cancer (PIN): A multicentre, randomised, controlled, phase 2 trial. EClinicalMedicine. 2022 Aug 11;52:101595. doi: 10.1016/j.eclinm.2022.101595. eCollection 2022 Oct. PMID 35990583
- [Background] Mekonnen N, Yang H, Shin YK. Homologous Recombination Deficiency in Ovarian, Breast, Colorectal, Pancreatic, Non-Small Cell Lung and Prostate Cancers, and the Mechanisms of Resistance to PARP Inhibitors. Front Oncol. 2022 Jun 17;12:880643. doi: 10.3389/fonc.2022.880643. eCollection 2022. PMID 35785170
- [Background] Valdiviezo, N. et al. MA12.04 FLAURA2: Impact of Tumor Burden on Outcomes of 1L Osimertinib ± Chemotherapy in Patients with EGFR-mutated Advanced NSCLC. Journal of Thoracic Oncology 19, S102 (2024)
- [Background] Yang, J. C. et al. MA12.03 FLAURA2: Resistance, and Impact of Baseline TP53 Alterations in Patients Treated With 1L Osimertinib ± Platinum-Pemetrexed. Journal of Thoracic Oncology 19, S101-S102 (2024)
- [Background] Planchard, D. et al. 512MO FLAURA2: Safety and CNS outcomes of first-line (1L) osimertinib (osi) ± chemotherapy (CTx) in EGFRm advanced NSCLC. Annals of Oncology 34, S1668 (2023)
- [Background] Cho BC, Lu S, Felip E, Spira AI, Girard N, Lee JS, Lee SH, Ostapenko Y, Danchaivijitr P, Liu B, Alip A, Korbenfeld E, Mourao Dias J, Besse B, Lee KH, Xiong H, How SH, Cheng Y, Chang GC, Yoshioka H, Yang JC, Thomas M, Nguyen D, Ou SI, Mukhedkar S, Prabhash K, D'Arcangelo M, Alatorre-Alexander J, Vazquez Limon JC, Alves S, Stroyakovskiy D, Peregudova M, Sendur MAN, Yazici O, Califano R, Gutierrez Calderon V, de Marinis F, Passaro A, Kim SW, Gadgeel SM, Xie J, Sun T, Martinez M, Ennis M, Fennema E, Daksh M, Millington D, Leconte I, Iwasawa R, Lorenzini P, Baig M, Shah S, Bauml JM, Shreeve SM, Sethi S, Knoblauch RE, Hayashi H; MARIPOSA Investigators. Amivantamab plus Lazertinib in Previously Untreated EGFR-Mutated Advanced NSCLC. N Engl J Med. 2024 Oct 24;391(16):1486-1498. doi: 10.1056/NEJMoa2403614. Epub 2024 Jun 26. PMID 38924756
- [Background] Planchard D, Janne PA, Cheng Y, Yang JC, Yanagitani N, Kim SW, Sugawara S, Yu Y, Fan Y, Geater SL, Laktionov K, Lee CK, Valdiviezo N, Ahmed S, Maurel JM, Andrasina I, Goldman J, Ghiorghiu D, Rukazenkov Y, Todd A, Kobayashi K; FLAURA2 Investigators. Osimertinib with or without Chemotherapy in EGFR-Mutated Advanced NSCLC. N Engl J Med. 2023 Nov 23;389(21):1935-1948. doi: 10.1056/NEJMoa2306434. Epub 2023 Nov 8. PMID 37937763
- [Background] Skoulidis F, Heymach JV. Co-occurring genomic alterations in non-small-cell lung cancer biology and therapy. Nat Rev Cancer. 2019 Sep;19(9):495-509. doi: 10.1038/s41568-019-0179-8. Epub 2019 Aug 12. PMID 31406302
- [Background] Hendriks LE, Kerr KM, Menis J, Mok TS, Nestle U, Passaro A, Peters S, Planchard D, Smit EF, Solomon BJ, Veronesi G, Reck M; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Oncogene-addicted metastatic non-small-cell lung cancer: ESMO Clinical Practice Guideline for diagnosis, treatment and follow-up. Ann Oncol. 2023 Apr;34(4):339-357. doi: 10.1016/j.annonc.2022.12.009. Epub 2023 Jan 23. No abstract available. PMID 36872130
- [Background] Oda K, Matsuoka Y, Funahashi A, Kitano H. A comprehensive pathway map of epidermal growth factor receptor signaling. Mol Syst Biol. 2005;1:2005.0010. doi: 10.1038/msb4100014. Epub 2005 May 25. PMID 16729045
- [Background] Hendriks LEL, Remon J, Faivre-Finn C, Garassino MC, Heymach JV, Kerr KM, Tan DSW, Veronesi G, Reck M. Non-small-cell lung cancer. Nat Rev Dis Primers. 2024 Sep 26;10(1):71. doi: 10.1038/s41572-024-00551-9. PMID 39327441
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751

DOCUMENTS (1):
  • Study Protocol (2025-09-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT07303218/Prot_000.pdf